CLINICAL TRIAL: NCT02868034
Title: Optimization of Spinal Manipulation Therapy (SMT) Protocols
Brief Title: Optimization of Spinal Manipulative Therapy Protocols
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Principal Investigator, Julie Fritz, Professor, University of Utah
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 1UH3AT009293-01 (NIH)
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-04

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Spinal Manipulation; Exercise
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- SMT Only (Experimental): Patients receive 2 sessions on SMT during week 1, no additional treatment.
  Interventions: Behavioral: SMT
- SMT extended (Experimental): 2 sessions of SMT in week 1 and 6 additional sessions of SMT during weeks 2-4.
  Interventions: Behavioral: SMT; Behavioral: SMT extended
- SMT with Activation Exercises (Experimental): 2 sessions of SMT during week 1 and 6 additional sessions of lumbar multifidus activating exercises during weeks 2-4.
  Interventions: Behavioral: SMT; Behavioral: Activation Exercises
- SMT with Mobilizing Exercises (Experimental): 2 sessions of SMT during week 1; 6 sessions of spinal mobilizing exercises during weeks 2-4.
  Interventions: Behavioral: SMT; Behavioral: Mobilizing Exercises
- SMT with Mobilizing and Activation Exercises (Experimental): 2 sessions of SMT during week 1; 6 sessions of lumbar multifidus activating exercises and spinal mobilizing exercises during weeks 2-4.
  Interventions: Behavioral: SMT; Behavioral: Mobilizing Exercises; Behavioral: Activation Exercises
- SMT extended with Mobilizing Exercises (Experimental): 2 sessions of SMT during week 1; 6 sessions of SMT and spinal mobilizing exercises during weeks 2-4.
  Interventions: Behavioral: SMT; Behavioral: Mobilizing Exercises; Behavioral: SMT extended
- SMT extended with Activation Exercises (Experimental): 2 sessions of SMT during week 1; 6 sessions of SMT and lumbar multifidus activating exercises during weeks 2-4.
  Interventions: Behavioral: SMT; Behavioral: Activation Exercises; Behavioral: SMT extended
- SMT extended with Activation and Mobilizing Exercises (Experimental): 2 sessions of SMT during week 1; 6 sessions of SMT, multifidus activating and spinal mobilizing exercises during weeks 2-4.
  Interventions: Behavioral: SMT; Behavioral: Mobilizing Exercises; Behavioral: Activation Exercises; Behavioral: SMT extended

INTERVENTIONS:
Behavioral: SMT — All patients receive 2 SMT sessions in the first week. The subject is supine. The clinician stands opposite the side to be manipulated and side-bends the subject away from the side to manipulate. The side to be manipulated is the more painful. If the subject cannot identify a more painful side the clinician selects a side. The clinician rotates the subject, and delivers a high-velocity, low-amplitude (HVLA) thrust to the pelvis in a posterior/inferior direction. The clinician notes if a cavitation (ie, a "pop") occurred. If it does, SMT treatment is complete. If no cavitation occurs, the subject is repositioned and SMT is performed again. If no cavitation occurs on the second attempt, the clinician manipulates the opposite side. A maximum of 2 attempts per side is permitted. If no cavitation is noted by that time, SMT treatment is complete. Substitution with a side-posture HVLA technique is allowed if the preferred technique is not possible due to subject preference or comfort.
  Other Names: Spinal Manipulative Therapy
Behavioral: Mobilizing Exercises — Mobilizing exercises will include a program of repeated movements progressing into end-ranges of spinal flexion and/or extension shown in past studies to improve ROM and reduce spinal stiffness. Patients will be instructed in mid-range exercises and will be further assessed for a directional preference. A directional preference is present if movement in a particular direction decreases LBP intensity or causes symptoms to centralize towards the midline. If a subject has a directional preference he or she will be prescribed exercises specifically in that direction along with mid-range exercise. Otherwise the subject will be assigned exercises moving into either flexion or extension based on the clinician's discretion. Subjects will perform their prescribed exercises at treatment sessions and will be instructed to perform the exercises daily on other days.
  Arms: SMT extended with Activation and Mobilizing Exercises; SMT extended with Mobilizing Exercises; SMT with Mobilizing Exercises; SMT with Mobilizing and Activation Exercises
Behavioral: Activation Exercises — Activation exercises are designed to facilitate use of the lumbar multifidus muscle. Exercises will begin with isometric multifidus contractions in different positions with clinician feedback and exercises to isometrically co-contract the multifidus and deep abdominal muscles. Subjects will also perform lumbar extensor strengthening exercises shown to produce 20%-50% of multifidus maximum voluntary contraction. Subjects will continue to perform isometric exercises throughout treatment. Subjects will perform their prescribed exercises at treatment sessions and will be instructed to perform the exercises daily on other days.
  Arms: SMT extended with Activation Exercises; SMT extended with Activation and Mobilizing Exercises; SMT with Activation Exercises; SMT with Mobilizing and Activation Exercises
Behavioral: SMT extended — This treatment involves 6 additional SMT sessions. Each SMT session is conducted as described previously.
  Arms: SMT extended; SMT extended with Activation Exercises; SMT extended with Activation and Mobilizing Exercises; SMT extended with Mobilizing Exercises

SUMMARY:
Research on spinal manipulative therapy for individuals with low back pain has been hampered by a lack of understanding of which of the physiologic effects produced by spinal manipulation are related to clinical benefit, and how these effects can be used to optimize treatment outcomes. Prior research has identified physiologic effects that relate to the clinical benefits from spinal manipulation treatment. The goal of this project is to examine strategies to use these effects to identify optimized treatment protocols. The results of this project will provide critical information for future clinical trials related to spinal manipulation.

DETAILED DESCRIPTION:
Low back pain (LBP) is a common and costly condition. Spinal manipulative therapy (SMT) is a common mind body intervention for individuals with LBP. Although SMT for LBP has been examined in numerous clinical studies, the literature on SMT remains unclear and even contradictory as to the effectiveness of this treatment. Studies that have supported SMT have generally found relatively small treatment effects. Many reasons have been offered for the inconsistent research literature and small effect sizes of SMT. A primary rationale offered is that the SMT protocols used in clinical research are not optimal, primarily due to a lack of understanding of the underlying mechanisms explaining the clinical benefits of SMT realized by some patients with LBP.

The prior work of this research team has identified two mechanisms explaining the therapeutic effects of SMT. These effects are a reduction in spinal stiffness and improved activation of the lumbar multifidus muscle. This research has also developed accurate, non-invasive methods to measure these effects and their response to SMT. The model identifying these two mechanisms has been validated in a second patient sample.

The overall goal of this proposal is to optimize SMT treatment protocols for patients with LBP. The optimization strategy in this study will evaluate SMT combined with other treatments known to modulate the same signals that underlie the clinical effects of SMT assessing both mechanistic (stiffness, lumbar multifidus activation) and patient-centered (function and pain) outcomes. This project will use innovative methodology to efficiently evaluate the effects of various individual treatment components towards an overall effect; identifying which components are contributing to the target outcomes and which, if any, may be discarded. All participants will be provided 2 sessions of SMT, and then will be randomized to a treatment group for an additional 3 weeks using a factorial design and stratified by responder status in order to evaluate different combinations of intervention components (muscle activation exercise, spinal mobilizing exercise, additional SMT) that work on the same pathways that modulate the same effects (spinal stiffness and muscle activation). Outcomes will include spinal stiffness and muscle activation measures as well as patient-reported outcomes assessed at baseline, and after 1 week, 4 weeks and 3 months. Results of this project will provide optimized SMT protocols that will be ready for application in future randomized controlled trials examining the efficacy and effectiveness of SMT.

ELIGIBILITY:
Inclusion Criteria:

I. Pain between the 12th rib and buttocks with or without symptoms into one or both legs, which, in the opinion of the examiner, originate from the lumbar region.

II. Age 18 - 60 years

III. Oswestry disability score > 20%

Exclusion Criteria:

I. Prior surgery to the lumbosacral spine

II. Currently pregnant

III. Currently receiving mind-body or exercise treatment for LBP from a healthcare provider (e.g., chiropractic, physical therapy, massage therapy, etc.)

IV. Neurogenic signs including any of the following: positive ipsi- or contra-lateral straight leg raise test; reflex, sensory, or strength deficit in a pattern consistent with lumbar nerve root compression

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 273 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2019-01-12 (Actual); Study Completion 2019-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Fritz, PhD, PT, Principal Investigator — University of Utah
Locations (2):
- University of Utah, Department of Physical Therapy, Salt Lake City, Utah, United States
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Fritz JM, Sharpe JA, Lane E, Santillo D, Greene T, Kawchuk G. Optimizing treatment protocols for spinal manipulative therapy: study protocol for a randomized trial. Trials. 2018 Jun 4;19(1):306. doi: 10.1186/s13063-018-2692-6. PMID 29866131

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled into Phase I of the study (enrollment - 1 week). After the completion of Phase I participants were randomized to an intervention arm for Phase II (1 week - 12 weeks). Baseline data are provided from the 1-week assessment, which corresponds to the time of randomization and beginning of Phase II.
Groups:
- Phase II - SMT Only: Patients receive 2 sessions on SMT during treatment Phase I, no additional treatment in Phase II.
  SMT: All patients receive 2 SMT sessions in the first week. The subject is supine. The clinician stands opposite the side to be manipulated and side-bends the subject away from the side to manipulate. The side to be manipulated is the more painful. If the subject cannot identify a more painful side the clinician selects a side. The clinician rotates the subject, and delivers a high-velocity, low-amplitude (HVLA) thrust to the pelvis in a posterior/inferior direction. The clinician notes if a cavitation (ie, a "pop") occurred. If it does, SMT treatment is complete. If no cavitation occurs, the subject is repositioned and SMT is performed again. If no cavitation occurs on the second attempt, the clinician manipulates the opposite side. A maximum of 2 attempts per side is permitted. If no cavitation is noted by that time, SMT treatment is complete. Substitution with a side-posture HVLA technique is allowed if the preferred technique is not possible due to subject preference or comfort.
- Phase II - SMT Extended: Patients received 2 sessions of SMT in during Phase I, and 6 additional sessions of SMT during Phase II.
  SMT: All patients receive 2 SMT sessions in the first week. The subject is supine. The clinician stands opposite the side to be manipulated and side-bends the subject away from the side to manipulate. The side to be manipulated is the more painful. If the subject cannot identify a more painful side the clinician selects a side. The clinician rotates the subject, and delivers a high-velocity, low-amplitude (HVLA) thrust to the pelvis in a posterior/inferior direction. The clinician notes if a cavitation (ie, a "pop") occurred. If it does, SMT treatment is complete. If no cavitation occurs, the subject is repositioned and SMT is performed again. If no cavitation occurs on the second attempt, the clinician manipulates the opposite side. A maximum of 2 attempts per side is permitted. If no cavitation is noted by that time, SMT treatment is complete. Substitution with a side-posture HVLA technique is allowed if the preferred technique is not possible due to subject preference or comfort.
  SMT extended: This treatment involves 6 additional SMT sessions. Each SMT session is conducted as described previously.
- Phase II - SMT With Activation Exercises: Patients received 2 sessions of SMT during Phase I, and 6 additional sessions of lumbar multifidus activating exercises during Phase II.
  SMT: All patients receive 2 SMT sessions in the first week. The subject is supine. The clinician stands opposite the side to be manipulated and side-bends the subject away from the side to manipulate. The side to be manipulated is the more painful. The clinician rotates the subject, and delivers a high-velocity, low-amplitude (HVLA) thrust to the pelvis in a posterior/inferior direction. Substitution with a side-posture HVLA technique is allowed.
  Activation Exercises: Activation exercises are designed to facilitate use of the lumbar multifidus muscle. Exercises will begin with isometric multifidus contractions in different positions with clinician feedback and exercises to isometrically co-contract the multifidus and deep abdominal muscles. Subjects will also perform lumbar extensor strengthening exercises shown to produce 20%-50% of multifidus maximum voluntary contraction. Subjects will continue to perform isometric exercises throughout treatment. Subjects will perform their prescribed exercises at treatment sessions and will be instructed to perform the exercises daily on other days.
- Phase II - SMT With Mobilizing Exercises: patients received 2 sessions of SMT during Phase I; and 6 sessions of spinal mobilizing exercises during Phase II.
  SMT: All patients receive 2 SMT sessions in the first week. The subject is supine. The clinician stands opposite the side to be manipulated and side-bends the subject away from the side to manipulate. The side to be manipulated is the more painful. The clinician rotates the subject, and delivers a high-velocity, low-amplitude (HVLA) thrust to the pelvis in a posterior/inferior direction. Substitution with a side-posture HVLA technique is allowed.
  Mobilizing Exercises: Mobilizing exercises will include a program of repeated movements progressing into end-ranges of spinal flexion and/or extension shown in past studies to improve ROM and reduce spinal stiffness. Patients will be instructed in mid-range exercises and will be further assessed for a directional preference. A directional preference is present if movement in a particular direction decreases LBP intensity or causes symptoms to centralize towards the midline. If a subject has a directional preference he or she will be prescribed exercises specifically in that direction along with mid-range exercise. Otherwise the subject will be assigned exercises moving into either flexion or extension based on the clinician's discretion. Subjects will perform their prescribed exercises at treatment sessions and will be instructed to perform the exercises daily on other days.
- Phase II - SMT With Mobilizing and Activation Exercises: Patients received 2 sessions of SMT during Phase I; and 6 sessions of lumbar multifidus activating exercises and spinal mobilizing exercises during Phase II.
  SMT: All patients receive 2 SMT sessions in the first week. The subject is supine. The clinician stands opposite the side to be manipulated and side-bends the subject away from the side to manipulate. The side to be manipulated is the more painful. The clinician rotates the subject, and delivers a high-velocity, low-amplitude (HVLA) thrust to the pelvis in a posterior/inferior direction. Substitution with a side-posture HVLA technique is allowed.
  Mobilizing Exercises: Mobilizing exercises include repeated movements in spinal flexion and/or extension. Patients will be instructed in mid-range exercises. If a subject has a directional preference he or she will be prescribed exercises specifically in that direction. Otherwise the subject will be assigned exercises moving into flexion or extension based on the clinician's discretion. Subjects will perform their prescribed exercises at treatment sessions and daily on other days.
  Activation Exercises: Activation exercises facilitate the lumbar multifidus muscle. Exercises begin with isometric multifidus contractions in different positions and co-contraction of multifidus and abdominals. Subjects also perform extensor strengthening exercises. Subjects will perform their prescribed exercises at treatment sessions daily on other days.
- Phase II - SMT Extended With Mobilizing Exercises: Patients received 2 sessions of SMT during Phase I; and 6 sessions of SMT and spinal mobilizing exercises during Phase II.
  SMT: All patients receive 2 SMT sessions in the first week. The subject is supine. The clinician stands opposite the side to be manipulated and side-bends the subject away from the side to manipulate. The side to be manipulated is the more painful. The clinician rotates the subject, and delivers a high-velocity, low-amplitude (HVLA) thrust to the pelvis in a posterior/inferior direction. Substitution with a side-posture HVLA technique is allowed.
  Mobilizing Exercises: Mobilizing exercises include repeated movements progressing into end-ranges of spinal flexion and/or extension. Patients will be instructed in mid-range exercises and are assessed for a directional preference. If a subject has a directional preference he or she will be prescribed exercises specifically in that direction along with mid-range exercise. Otherwise the subject will be assigned exercises moving into either flexion or extension based on the clinician's discretion. Subjects will perform their prescribed exercises at treatment sessions and will be instructed to perform the exercises daily on other days.
  SMT extended: This treatment involves 6 additional SMT sessions. Each SMT session is conducted as described previously.
- Phase II - SMT Extended With Activation Exercises: Patients received 2 sessions of SMT during Phase I; and 6 sessions of SMT and lumbar multifidus activating exercises during Phase II.
  SMT: All patients receive 2 SMT sessions in the first week. The subject is supine. The clinician stands opposite the side to be manipulated and side-bends the subject away from the side to manipulate. The side to be manipulated is the more painful. The clinician rotates the subject, and delivers a high-velocity, low-amplitude (HVLA) thrust to the pelvis in a posterior/inferior direction. Substitution with a side-posture HVLA technique is allowed.
  Activation Exercises: Activation exercises are designed to facilitate use of the lumbar multifidus muscle. Exercises will begin with isometric multifidus contractions in different positions with clinician feedback and exercises to isometrically co-contract the multifidus and deep abdominal muscles. Subjects will also perform lumbar extensor strengthening exercises shown to produce 20%-50% of multifidus maximum voluntary contraction. Subjects will continue to perform isometric exercises throughout treatment. Subjects will perform their prescribed exercises at treatment sessions and will be instructed to perform the exercises daily on other days.
  SMT extended: This treatment involves 6 additional SMT sessions. Each SMT session is conducted as described previously.
- Phase II - SMT Extended With Activation and Mobilizing Exercises: Patients received 2 sessions of SMT during Phase I; and 6 sessions of SMT, multifidus activating and spinal mobilizing exercises during Phase II.
  SMT: All patients receive 2 SMT sessions in the first week. The subject is supine. The clinician stands opposite the side to be manipulated and side-bends the subject away from the side. The side to be manipulated is the more painful. The clinician rotates the subject, and delivers a high-velocity, low-amplitude (HVLA) thrust to the pelvis in a posterior/inferior direction. Substitution with a side-posture HVLA technique is allowed.
  Mobilizing Exercises: include repeated movements in spinal flexion and/or extension. Patients will be instructed in mid-range exercises. If a subject has a directional preference he or she will be prescribed exercises specifically in that direction. Otherwise the subject will be assigned exercises moving into flexion or extension based on the clinician's discretion. Subjects will perform their prescribed exercises at treatment sessions and daily on other days.
  Activation Exercises: Activation exercises facilitate the lumbar multifidus muscle. Exercises begin with isometric multifidus contractions in different positions and co-contraction of multifidus and abdominals. Subjects also perform extensor strengthening exercises. Subjects will perform their prescribed exercises at treatment sessions daily on other days.
  SMT extended: 6 additional SMT sessions, each conducted as described previously.
Period: Overall Study
Arm/Group | Phase II - SMT Only | Phase II - SMT Extended | Phase II - SMT With Activation Exercises | Phase II - SMT With Mobilizing Exercises | Phase II - SMT With Mobilizing and Activation Exercises | Phase II - SMT Extended With Mobilizing Exercises | Phase II - SMT Extended With Activation Exercises | Phase II - SMT Extended With Activation and Mobilizing Exercises
Started | 30 | 29 | 30 | 31 | 30 | 29 | 30 | 32
Completed | 22 | 23 | 26 | 27 | 24 | 26 | 24 | 26
Not Completed | 8 | 6 | 4 | 4 | 6 | 3 | 6 | 6

BASELINE CHARACTERISTICS:
Population: 315 individuals provided consent and 273 met all eligibility criteria and enrolled in Phase I. Of these 32 (11.7%) withdrew during treatment phase I, leaving 241 participants who completed the 1-week assessment and were randomized to receive additional treatment components in Phase II. The Phase II baseline information is provided.
Groups:
- Phase II - No Further Treatment: Phase II baseline values from the 1-weekassessment for participants who did not receive additional treatment in Phase II
- Phase II - Extended SMT Only: Phase II baseline values from the 1-weekassessment for participants who received 2 sessions per week of additional SMT in Phase II
- Phase II - Activating Exercise Component Only: Phase II baseline values from the 1-weekassessment for participants who received 2 sessions per week of activating exercises only in Phase II
- Phase II - Mobilizing Exercise Component Only: Phase II baseline values from the 1-weekassessment for participants who received 2 sessions per week of mobilizing exercises only in Phase II
- Phase II i SMT and Activating Exercise Component: Phase II baseline values from the 1-weekassessment for participants who received 2 sessions per week of activating exercises and SMT in Phase II
- Phase II - - SMT With Mobilizing Exercise Component: Phase II baseline values from the 1-weekassessment for participants who received 2 sessions per week of mobilizing exercises and SMT in Phase II
- Phase II - Activating Exercise and Mobilizing Exercise Components: Phase II baseline values from the 1-weekassessment for participants who received 2 sessions per week of mobilizing exercises and activating exercises in Phase II
- Phase II - SMT With Mobilizing Exercise and Activating Exercise: Phase II baseline values from the 1-weekassessment for participants who received 2 sessions per week of mobilizing exercises and activating exercises and SMT in Phase II
- Total: Total of all reporting groups
Arm/Group | Phase II - No Further Treatment | Phase II - Extended SMT Only | Phase II - Activating Exercise Component Only | Phase II - Mobilizing Exercise Component Only | Phase II i SMT and Activating Exercise Component | Phase II - - SMT With Mobilizing Exercise Component | Phase II - Activating Exercise and Mobilizing Exercise Components | Phase II - SMT With Mobilizing Exercise and Activating Exercise | Total
Number analyzed (Participants) | 30 | 29 | 30 | 31 | 30 | 29 | 30 | 32 | 241
Age, Continuous [Mean (Standard Deviation); unit: years] — Data represents the Phase II baseline data per treatment group. Population: A total of 273 met all eligibility criteria and enrolled in Phase I of the study. Of these 32 (11.7%) withdrew during treatment phase I, leaving 241 participants who completed the 1-week assessment and were randomized to receive additional treatment components in Phase II.
  years
    Phase II baseline age | 42.6 (11.5) | 36.3 (9.8) | 41.1 (12.6) | 38.1 (10.5) | 41.2 (13.7) | 40.4 (12) | 40.5 (10.5) | 38.8 (12.3) | 39.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Measure Description: Data represents the Phase II baseline data per treatment group.
  Participants
    Phase II - Baseline Sex: Female | 18 | 20 | 20 | 19 | 18 | 15 | 16 | 18 | 144
    Phase II - Baseline Sex: Male | 12 | 9 | 10 | 12 | 12 | 14 | 14 | 14 | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Measure Description: Measure Description: Data represents the Phase II baseline data per treatment group.
  Participants
    Hispanic or Latino | 1 | 3 | 4 | 3 | 3 | 6 | 0 | 0 | 20
    Not Hispanic or Latino | 28 | 25 | 26 | 28 | 27 | 21 | 30 | 32 | 217
    Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Measure Description: Measure Description: Data represents the Phase II baseline data per treatment group.
  Participants
    American Indian or Alaska Native | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
    Asian | 2 | 3 | 5 | 4 | 2 | 2 | 3 | 4 | 25
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 7
    White | 22 | 19 | 19 | 21 | 24 | 21 | 25 | 25 | 176
    More than one race | 1 | 1 | 2 | 3 | 2 | 2 | 0 | 2 | 13
    Unknown or Not Reported | 1 | 5 | 3 | 3 | 1 | 3 | 0 | 0 | 16
Chronic LBP [Count of Participants; unit: Participants] — Data represents the Phase II baseline data per treatment group.
  Measure Description: Chronic back pain defined as participants reporting the duration of their current low back symptoms was greater than 3 months.
  Participants | 24 | 22 | 23 | 25 | 26 | 20 | 21 | 22 | 183
Oswestry [Mean (Standard Deviation); unit: units on a scale] — Measure Description: Data represents the Phase II baseline data per treatment group.
  units on a scale | 35.7 (11.8) | 36.1 (17.7) | 33.9 (10.0) | 30.6 (8.6) | 36.3 (11.5) | 29.1 (9.5) | 32.7 (9.3) | 38.6 (12.0) | 34.4 (11.8)
Pain intensity [Mean (Standard Deviation); unit: units on a scale] — Data represents the Phase II baseline data per treatment group.
  units on a scale | 4.4 (1.5) | 4.9 (2.0) | 4.8 (1.5) | 4.4 (1.7) | 4.5 (1.5) | 4.4 (1.7) | 4.5 (1.6) | 4.9 (1.7) | 4.6 (1.7)
Multifidus Activation [Mean (Standard Deviation); unit: percentage increase in thickness] — Data represents the Phase II baseline data per treatment group.
  Measure Description: Percentage increase in thickness of the multifidus muscle assessed using ultrasound comparing the muscle at rest versus submaximal contraction. Higher values indicate greater muscle activation.
  percentage increase in thickness | 11.4 (9.5) | 9.5 (9.4) | 13.6 (11.4) | 11.6 (8.5) | 14.2 (10.9) | 10.7 (9.1) | 10.0 (8.9) | 11.6 (8.2) | 11.2 (9.3)
Spinal Stiffness [Mean (Standard Deviation); unit: N/mm] — Data represents the Phase II baseline data per treatment group.
  Measure Description: Spinal stiffness is assessed with the VerteTrack device that applies a vertical load along the lumbar spine of a prone participant. The indenter houses a sensor to provide continuous, real-time quantification of spinal deformation in response to a defined load. Stiffness was determined as the ratio of the maximum applied force to the resultant displacement in N/mm. Higher numbers indicate greater amounts of stiffness.
  N/mm | 6.0 (1.2) | 5.8 (1.4) | 5.9 (1.3) | 6.3 (1.1) | 5.7 (1.2) | 5.9 (1.4) | 5.7 (1.1) | 5.9 (1.0) | 6.0 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Spinal Stiffness
Description: Spinal stiffness is assessed with the VerteTrack device that applies a vertical load along the lumbar spine of a prone participant. The indenter houses a sensor to provide continuous, real-time quantification of spinal deformation in response to a defined load. Stiffness was determined as the ratio of the maximum applied force to the resultant displacement in N/mm. Higher numbers indicate greater amounts of stiffness.
Time Frame: Assessed at Phase II Baseline, 4 weeks, 12 weeks. 4 weeks and 12 weeks reported. Phase II baseline values were constrained to be equal to a common overall mean for analyses.
Population: Results were examined based on the main effects and interactions among the 3 treatment components in the factorial study design (SMT, Mobilizing Exercise, Activating Exercise). Scores were missing for participants in the SMT group (n=21 at 4 weeks and 12 weeks), Mobilizing exercise (n=14 at 4 weeks and n=19 at 12 weeks), and Activating exercise (n=16 at 4 weeks and n=22 at 12 weeks)
Measure: Mean (97.5% Confidence Interval); unit: N/mm
Groups:
- SMT Treatment Component: Participants who received extended SMT in weeks 2-4 based on randomized assignment in the factorial study design.
- Mobilizing Exercise Component: Participants who received mobilizing exercises in weeks 2-4 based on randomized assignment in the factorial study design.
- Activating Exercise Component: Participants who received activating exercises in weeks 2-4 based on randomized assignment in the factorial study design.
Arm/Group | SMT Treatment Component | Mobilizing Exercise Component | Activating Exercise Component
Number analyzed (Participants) | 99 | 108 | 106
N/mm
  Spinal Stiffness measure at 4 weeks | 6.20 [5.98 to 6.41] | 6.28 [6.07 to 6.48] | 6.10 [5.90 to 6.31]
  Spinal Stiffness measure at 12 weeks: number analyzed (Participants) | 99 | 103 | 100
  Spinal Stiffness measure at 12 weeks | 6.07 [5.85 to 6.28] | 6.16 [5.96 to 6.37] | 6.06 [5.85 to 6.27]
Statistical Analysis 1: Comparison: SMT Treatment Component; SMT Component Main Effects at 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; Consistent with the randomized design, mean values for the Phase II baseline were constrained to be equal to a common overall mean; Mean Difference (Final Values) = -0.02, 97.5% CI 2-sided [-0.26 to 0.22] — A negative value indicates greater reduction in stiffness when the component was used
Statistical Analysis 2: Comparison: SMT Treatment Component; SMT Component Main Effects after 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.17, 97.5% CI 2-sided [-0.43 to 0.09] — A negative value indicates greater reduction in stiffness when the component was used
Statistical Analysis 3: Comparison: Mobilizing Exercise Component; Mobilizing Exercise Treatment Component Main Effects at 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.14, 97.5% CI 2-sided [-0.11 to 0.38] — A negative value indicates greater reduction in stiffness when the component was used
Statistical Analysis 4: Comparison: Mobilizing Exercise Component; Mobilizing Exercise Component Main Effects at 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.03, 97.5% CI 2-sided [-0.23 to 0.29] — A negative value indicates greater reduction in stiffness when the component was used
Statistical Analysis 5: Comparison: Activating Exercise Component; Activating Exercise Component Main Effect at 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.20, 97.5% CI 2-sided [-0.45 to 0.04] — A negative value indicates greater reduction in stiffness when the component was used
Statistical Analysis 6: Comparison: Activating Exercise Component; Activating Exercise Component Main Effect at 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.19, 97.5% CI 2-sided [-0.45 to 0.07] — A negative value indicates greater change when the component was used
Statistical Analysis 7: Comparison: Mobilizing Exercise Component vs Activating Exercise Component; Pairwise interaction effect of mobilizing and activating exercise components after 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = -0.17, 97.5% CI 2-sided [-0.66 to 0.32]
Statistical Analysis 8: Comparison: Mobilizing Exercise Component vs Activating Exercise Component; Pairwise interaction effect of mobilizing and activating exercise components after 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = -0.10, 97.5% CI 2-sided [-0.62 to 0.42]
Statistical Analysis 9: Comparison: SMT Treatment Component vs Activating Exercise Component; Pairwise interaction effect of SMT and activating exercise components after 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = 0.13, 97.5% CI 2-sided [-0.36 to 0.62]
Statistical Analysis 10: Comparison: SMT Treatment Component vs Activating Exercise Component; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = 0.50, 97.5% CI 2-sided [-0.02 to 1.02]
Statistical Analysis 11: Comparison: SMT Treatment Component vs Mobilizing Exercise Component; Pairwise interaction effect of SMT and mobilizing exercise components after 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = -0.17, 97.5% CI 2-sided [-0.66 to 0.32]
Statistical Analysis 12: Comparison: SMT Treatment Component vs Mobilizing Exercise Component; Pairwise interaction effect of SMT and mobilizing exercise components after 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = 0.39, 97.5% CI 2-sided [-0.13 to 0.91]
Statistical Analysis 13: Comparison: SMT Treatment Component vs Mobilizing Exercise Component vs Activating Exercise Component; Three-way interaction effect of SMT, activating exercise and mobilizing exercise components after 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; 3-way interaction relative mean dif. = 0.25, 97.5% CI 2-sided [-0.24 to 0.74]
Statistical Analysis 14: Comparison: SMT Treatment Component vs Mobilizing Exercise Component vs Activating Exercise Component; Three-way interaction effect of SMT, activating exercise and mobilizing exercise components after 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; 3-way interaction relative mean dif. = 0.40, 97.5% CI 2-sided [-0.12 to 0.92]

2. Primary Outcome: Multifidus Activation
Description: Multifidus activation was measured with brightness-mode ultrasound images using a 60mm, 2-5 MHz curvilinear array. Images are acquired with the multifidus at rest and during submaximal contraction. Three images in each state are acquired and averaged. Muscle activation is calculated as the change in thickness at rest and submaximal contraction and expressed as a percentage change. Greater numbers indicate higher muscle activation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (97.5% Confidence Interval); unit: percentage
Arm/Group | SMT Treatment Component | Mobilizing Exercise Component | Activating Exercise Component
Number analyzed (Participants) | 99 | 108 | 106
percentage
  Multifidus Activation 4 weeks | 12.10 [10.20 to 14.0] | 12.42 [10.56 to 14.28] | 12.0 [10.09 to 13.84]
  Multifidus Activation 12 weeks: number analyzed (Participants) | 99 | 103 | 106
  Multifidus Activation 12 weeks | 12.20 [10.28 to 14.12] | 12.74 [10.87 to 14.62] | 12.10 [10.22 to 13.97]
Statistical Analysis 1: Comparison: SMT Treatment Component; SMT Component Main Effects at 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.57, 97.5% CI 2-sided [-2.67 to 1.52]; A positive value indicates greater improvement in muscle activation when the component was used
Statistical Analysis 2: Comparison: SMT Treatment Component; SMT Component Main Effects at 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.37, 97.5% CI 2-sided [-2.76 to 2.02] — A positive value indicates greater improvement in muscle activation when the component was used
Statistical Analysis 3: Comparison: Mobilizing Exercise Component; Mobilizing Component Main Effects at 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.06, 97.5% CI 2-sided [-2.03 to 2.16] — A positive value indicates greater improvement in muscle activation when the component was used
Statistical Analysis 4: Comparison: Mobilizing Exercise Component; Mobilizing Component Main Effects at 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.71, 97.5% CI 2-sided [-1.68 to 3.11] — A positive value indicates greater improvement in muscle activation when the component was used
Statistical Analysis 5: Comparison: Activating Exercise Component; Activating Exercise Component at 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.85, 97.5% CI 2-sided [-2.94 to 1.25] — A positive value indicates greater improvement in muscle activation when the component was used
Statistical Analysis 6: Comparison: Activating Exercise Component; Activating Exercise Component at 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.57, 97.5% CI 2-sided [-2.97 to 1.82] — A positive value indicates greater improvement in muscle activation when the component was used
Statistical Analysis 7: Comparison: Mobilizing Exercise Component vs Activating Exercise Component; Pairwise interaction effect of mobilizing and activating exercise components after 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = 0.80, 97.5% CI 2-sided [-3.39 to 4.99]
Statistical Analysis 8: Comparison: Mobilizing Exercise Component vs Activating Exercise Component; Pairwise interaction effect of mobilizing and activating exercise components after 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = -0.68, 97.5% CI 2-sided [-5.47 to 4.11]
Statistical Analysis 9: Comparison: SMT Treatment Component vs Activating Exercise Component; Pairwise interaction effect of SMT and activating exercise components after 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = -1.56, 97.5% CI 2-sided [-5.75 to 2.63]
Statistical Analysis 10: Comparison: SMT Treatment Component vs Activating Exercise Component; Pairwise interaction effect of SMT and activating exercise components after 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = 1.42, 97.5% CI 2-sided [-3.37 to 6.21]
Statistical Analysis 11: Comparison: SMT Treatment Component vs Mobilizing Exercise Component; Pairwise interaction effect of SMT and mobilizing exercise components after 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = -0.44, 97.5% CI 2-sided [-4.63 to 3.75]
Statistical Analysis 12: Comparison: SMT Treatment Component vs Mobilizing Exercise Component; Pairwise interaction effect of SMT and mobilizing exercise components after 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = 2.01, 97.5% CI 2-sided [-2.77 to 6.80]
Statistical Analysis 13: Comparison: SMT Treatment Component vs Mobilizing Exercise Component vs Activating Exercise Component; Three-way interaction effect of SMT, activating exercise and mobilizing exercise components after 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; 3-way interaction relative mean dif. = -0.18, 97.5% CI 2-sided [-4.37 to 4.01]
Statistical Analysis 14: Comparison: SMT Treatment Component vs Mobilizing Exercise Component vs Activating Exercise Component; Three-way interaction effect of SMT, activating exercise and mobilizing exercise components after 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; 3-way interaction relative mean dif. = 0.56, 97.5% CI 2-sided [-4.22 to 5.35]

3. Secondary Outcome: Oswestry Disability Index
Description: The Oswestry Disability Index measures back pain-related disability. The scale contains 10 items with a minimum score of zero and maximum score of 100. Higher numbers indicate more disability. There are no subscales.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (97.5% Confidence Interval); unit: units on a scale
Arm/Group | SMT Treatment Component | Mobilizing Exercise Component | Activating Exercise Component
Number analyzed (Participants) | 99 | 108 | 106
units on a scale
  Oswestry 4 week outcomes | 21.74 [19.23 to 24.25] | 21.64 [19.18 to 24.1] | 21.15 [18.7 to 23.61]
  Oswestry 12 week outcomes: number analyzed (Participants) | 99 | 103 | 100
  Oswestry 12 week outcomes | 19.73 [17.05 to 22.42] | 18.97 [16.33 to 21.62] | 18.02 [15.38 to 20.66]
Statistical Analysis 1: Comparison: SMT Treatment Component; SMT Treatment Component Main Effect at 4-weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.16, 97.5% CI 2-sided [-4.0 to 1.68] — A negative value indicates greater improvement in disability when the component was used
Statistical Analysis 2: Comparison: SMT Treatment Component; SMT Treatment Component Main Effect at 12-weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.20, 97.5% CI 2-sided [-3.46 to 3.07] — A negative value indicates greater improvement in disability when the component was used
Statistical Analysis 3: Comparison: Mobilizing Exercise Component; Mobilizing Exercise Treatment Component main effect after 4-weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.36, 97.5% CI 2-sided [-4.2 to 1.48] — A negative value indicates greater improvement in disability when the component was used
Statistical Analysis 4: Comparison: Mobilizing Exercise Component; Mobilizing Exercise Treatment Component main effect after 12-weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.72, 97.5% CI 2-sided [-4.99 to 1.55] — A negative value indicates greater improvement in disability when the component was used
Statistical Analysis 5: Comparison: Activating Exercise Component; Activating Exercise Treatment Component main effect after 4-weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.34, 97.5% CI 2-sided [-5.18 to 0.50] — A negative value indicates greater improvement in disability when the component was used
Statistical Analysis 6: Comparison: Activating Exercise Component; Activating Treatment Component Main Effect after 12-weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.62, 97.5% CI 2-sided [-6.89 to -0.35] — A negative value indicates greater improvement in disability when the component was used
Statistical Analysis 7: Comparison: Mobilizing Exercise Component vs Activating Exercise Component; Pairwise interaction effect of mobilizing and activating exercise components after 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = 3.24, 97.5% CI 2-sided [-2.45 to 8.92]
Statistical Analysis 8: Comparison: Mobilizing Exercise Component vs Activating Exercise Component; Pairwise interaction effect of mobilizing and activating exercise components after 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = 4.34, 97.5% CI 2-sided [-2.19 to 10.87]
Statistical Analysis 9: Comparison: SMT Treatment Component vs Activating Exercise Component; Pairwise interaction effect of SMT and activating exercise components after 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = 0.57, 97.5% CI 2-sided [-5.12 to 6.25]
Statistical Analysis 10: Comparison: SMT Treatment Component vs Activating Exercise Component; Pairwise interaction effect of SMT and activating exercise components after 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = -0.67, 97.5% CI 2-sided [-7.20 to 5.87]
Statistical Analysis 11: Comparison: SMT Treatment Component vs Mobilizing Exercise Component; Pairwise interaction effect of SMT and mobilizing exercise components after 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = 4.64, 97.5% CI 2-sided [-1.04 to 10.32]
Statistical Analysis 12: Comparison: SMT Treatment Component vs Mobilizing Exercise Component; Pairwise interaction effect of SMT and mobilizing exercise components after 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = 1.49, 97.5% CI 2-sided [-5.04 to 8.02]
Statistical Analysis 13: Comparison: SMT Treatment Component vs Mobilizing Exercise Component vs Activating Exercise Component; 3-way interaction effect of SMT, activating exercise and mobilizing exercise components after 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; 3-way interaction relative mean dif. = -0.86, 97.5% CI 2-sided [-6.54 to 4.82]
Statistical Analysis 14: Comparison: SMT Treatment Component vs Mobilizing Exercise Component vs Activating Exercise Component; 3-way interaction effect of SMT, activating exercise and mobilizing exercise components after 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; 3-way interaction relative mean dif. = 0.04, 97.5% CI 2-sided [-6.50 to 6.57]

4. Secondary Outcome: Pain Intensity
Description: A 0-10 numeric pain rating is used to assess pain intensity. The minimum score is zero, maximum score is 10. Higher numbers indicate greater pain intensity. There are no subscales.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (97.5% Confidence Interval); unit: units on a scale
Arm/Group | SMT Treatment Component | Mobilizing Exercise Component | Activating Exercise Component
Number analyzed (Participants) | 99 | 108 | 106
units on a scale
  Pain intensity rating 4 weeks | 3.13 [2.76 to 3.51] | 2.98 [2.61 to 3.34] | 3.13 [2.76 to 3.49]
  Pain intensity rating 12 weeks: number analyzed (Participants) | 99 | 103 | 100
  Pain intensity rating 12 weeks | 3.10 [2.69 to 3.51] | 2.97 [2.56 to 3.37] | 2.96 [2.56 to 3.37]
Statistical Analysis 1: Comparison: SMT Treatment Component; SMT Treatment Component Main Effect at 4-weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.14, 97.5% CI 2-sided [-0.60 to 0.32] — A negative value indicates greater reduction in pain intensity when the component was used
Statistical Analysis 2: Comparison: SMT Treatment Component; SMT Treatment Component Main Effects at 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.08, 97.5% CI 2-sided [-0.44 to 0.61] — A negative value indicates greater reduction in pain intensity when the component was used
Statistical Analysis 3: Comparison: Mobilizing Exercise Component; Mobilizing Exercise Component Main Effects at 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.46, 97.5% CI 2-sided [-0.92 to 0.0] — A negative value indicates greater reduction in pain intensity when the component was used
Statistical Analysis 4: Comparison: Mobilizing Exercise Component; Mobilizing Exercise Component Main Effects at 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.18, 97.5% CI 2-sided [-0.70 to 0.34] — A negative value indicates greater reduction in pain intensity when the component was used
Statistical Analysis 5: Comparison: Activating Exercise Component; Activating Exercise Component Main Effects at 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.16, 97.5% CI 2-sided [-0.62 to 0.30] — A negative value indicates greater reduction in pain intensity when the component was used
Statistical Analysis 6: Comparison: Activating Exercise Component; Activating Exercise Component Main Effects at 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.19, 97.5% CI 2-sided [-0.71 to 0.33] — A negative value indicates greater reduction in pain intensity when the component was used
Statistical Analysis 7: Comparison: Mobilizing Exercise Component vs Activating Exercise Component; Pairwise interaction effect of mobilizing and activating exercise components after 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = 0.38, 97.5% CI 2-sided [-0.54 to 1.30]
Statistical Analysis 8: Comparison: Mobilizing Exercise Component vs Activating Exercise Component; Pairwise interaction effect of mobilizing and activating exercise components after 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = 0.45, 97.5% CI 2-sided [-0.60 to 1.49]
Statistical Analysis 9: Comparison: SMT Treatment Component vs Activating Exercise Component; Pairwise interaction effect of SMT and activating exercise components after 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = 0.12, 97.5% CI 2-sided [-0.80 to 1.04]
Statistical Analysis 10: Comparison: SMT Treatment Component vs Activating Exercise Component; Pairwise interaction effect of SMT and activating exercise components after 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = 0.23, 97.5% CI 2-sided [-0.81 to 1.28]
Statistical Analysis 11: Comparison: SMT Treatment Component vs Mobilizing Exercise Component; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = 0.89, 97.5% CI 2-sided [-0.03 to 1.81]
Statistical Analysis 12: Comparison: SMT Treatment Component vs Mobilizing Exercise Component; Pairwise interaction effect of SMT and mobilizing exercise components after 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; interaction relative mean difference = -0.02, 97.5% CI 2-sided [-1.07 to 1.02]
Statistical Analysis 13: Comparison: SMT Treatment Component vs Mobilizing Exercise Component vs Activating Exercise Component; 3-way interaction effect of SMT, activating exercise and mobilizing exercise components after 4 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; 3-way interaction relative mean dif. = 0.71, 97.5% CI 2-sided [-0.21 to 1.63]
Statistical Analysis 14: Comparison: SMT Treatment Component vs Mobilizing Exercise Component vs Activating Exercise Component; 3-way interaction effect of SMT, activating exercise and mobilizing exercise components after 12 weeks; Test type: Superiority; p = 0.025, Mixed Models Analysis; 3-way interaction relative mean dif. = 0.0, 97.5% CI 2-sided [-1.05 to 1.04]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 12 week period from baseline to final assessment including both Phase I and Phase II (post-randomization). Events reported by Phase II treatment group may have occurred at any point over the 12-week study period. Among the 32 participants who withdrew before randomization, 4 participants reported 5 adverse events. All events were an increase in symptoms of back pain, spasm or stiffness.
Groups:
- No Further Treatment: Participants received no additional treatment in weeks 2-4
- Extended SMT: Participants received 2 sessions per week of additional SMT in weeks 2-4
- Activating Exercise Component Only: Participants received activating exercises only in weeks 2-4.
- Mobilizing Exercise Component Only: Participants received mobilizing exercises only in weeks 2-4.
- SMT With Activating Exercise Component: Participants received SMT and activating exercises in weeks 2-4.
- SMT With Mobilizing Exercise Component: Participants received SMT and mobilizing exercises in weeks 2-4.
- Activating Exercise and Mobilizing Exercise Components: Participants received activating exercises and mobilizing exercises in weeks 2-4.
- SMT With Activating Exercise and Mobilizing Exercise Components: Participants received SMT with both activating exercises and mobilizing exercises in weeks 2-4.
Arm/Group | No Further Treatment | Extended SMT | Activating Exercise Component Only | Mobilizing Exercise Component Only | SMT With Activating Exercise Component | SMT With Mobilizing Exercise Component | Activating Exercise and Mobilizing Exercise Components | SMT With Activating Exercise and Mobilizing Exercise Components
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29 | 0/30 | 0/31 | 0/30 | 0/29 | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29 | 0/30 | 0/31 | 0/30 | 0/29 | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 3/30 | 8/29 | 9/30 | 10/31 | 12/30 | 7/29 | 5/30 | 13/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Further Treatment (N=30) | Extended SMT (N=29) | Activating Exercise Component Only (N=30) | Mobilizing Exercise Component Only (N=31) | SMT With Activating Exercise Component (N=30) | SMT With Mobilizing Exercise Component (N=29) | Activating Exercise and Mobilizing Exercise Components (N=30) | SMT With Activating Exercise and Mobilizing Exercise Components (N=32)
Increased low back symptoms from treatment (Musculoskeletal and connective tissue disorders) | 3 (4) | 7 (9) | 8 (14) | 10 (17) | 10 (15) | 7 (9) | 4 (7) | 12 (16) — Reported increase in low back pain, soreness, stiffness or spasm during or following a treatment session
Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) — Participants reporting motor vehicle accident or fall outside of treatment
Surgical procedures (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participants reporting a surgical procedure other than back surgery
Reinjured Low Back (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) — Reinjured low back attributable to an event outside of treatment session

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/34/NCT02868034/Prot_SAP_000.pdf